CLINICAL TRIAL: NCT01294163
Title: Efficacy and Safety of Xenon Anaesthesia Compared to Sevoflurane Anaesthesia and Total Intravenous Anaesthesia for On-pump Coronary Artery Bypass Graft Surgery: a Randomised, Three-arm, Single-blind, International Study
Brief Title: Xenon Compared to Sevoflurane and Total Intravenous Anaesthesia for Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALMED-09-C3-026
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease; General Anesthetic Drug Allergy; Coronary Artery Bypass Graft Surgery
Keywords: Xenon; Sevoflurane; Propofol; Total intravenous anaesthesia; Anaesthesia; Coronary artery disease; Coronary artery bypass graft
MeSH Terms: conditions — Coronary Artery Disease | interventions — Xenon; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xenon (Experimental)
  Interventions: Drug: Xenon
- Sevoflurane (Active Comparator)
  Interventions: Drug: Sevoflurane
- Total intravenous anaesthesia (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Xenon — Inhaled xenon, maximal inspired concentration of 65%.
  Arms: Xenon
Drug: Sevoflurane — Inhaled sevoflurane, maximal inspired concentration of 1.8%.
  Arms: Sevoflurane
Drug: Propofol — Hourly dose of 2-4 mg/kg
  Arms: Total intravenous anaesthesia

SUMMARY:
Xenon is a gaseous anaesthetic agent registered in several European countries. It has been administered safely during cardiac surgery in pilot studies. In animal studies, xenon decreases the size of experimental myocardial infarction.

This 3-arm study will compare xenon, sevoflurane and a propofol-based total intravenous anaesthesia for maintenance of anaesthesia during coronary artery bypass graft surgery conducted with extra-corporeal circulation. Xenon and sevoflurane will be administered before and after extracorporeal circulation. Propofol will be administered during extracorporeal circulation in the three groups of patients.

The study will compare the postoperative myocardial damage observed 24 hours after surgery from blood levels of troponin I, a largely accepted biomarker of myocardial necrosis. The main hypothesis is that the myocardial damage observed after xenon administration will not be superior to the damage observed after sevoflurane administration (non-inferiority). The second hypothesis is that the myocardial damage observed after xenon administration will be inferior to the damage observed after total intravenous anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* elective surgery, planned coronary artery bypass graft
* moderate hypothermia or normothermia
* cardiac arrest cold and warm cardioplegia
* normal of moderately impaired left ventricular systolic function
* written informed consent

Exclusion Criteria:

* pregnancy or child bearing potential
* ongoing treatment with nicorandil or sulfonylurea medication
* severe renal or hepatic dysfunction
* ongoing myocardial infarction or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan HOFLAND, MD, PhD, Principal Investigator — Thorax Centre Erasmus MC, Rotterdam, the Netherlands
Locations (17):
- France (8):
  - Hôpital Cardiovasculaire et Pneumologique Louis Pradel, Bron
  - CHU de Caen, Caen
  - Hôpital G&R Laennec - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalo-Universitaire Pitié-Salpetrière, Paris
  - Hôpital du Haut-Lévêque, Pessac
  - Hôpital Pontchaillou, Rennes
  - Hôpitaux Universitaires de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Centre Hospitalier de Rangueil, Toulouse
- Germany (6):
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - University Hospital Aachen, Aachen
  - Klinikum Links der Weser - Senator-Wessling-Str. 1, Bremen
  - University Hospital Frankfurt AM Main, Frankfurt
  - UniversitatsKlinikum Schleswig-Holstein, Lübeck
  - University Hospital ROSTOCK, Rostock
- Policlinico Umberto I, Rome, Italy
- Netherlands (2):
  - Academic Medical Center - University of Amsterdam, Amsterdam
  - Thorax Center - Erasmus MC, Rotterdam

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 542 patients were enrolled (509 met the inclusion criteria) from 17 centres in 4 countries; 8 sites in France, 6 sites in Germany, 1 site in Italy and 2 sites in The Netherlands.
  Date of first enrolment: 20 April 2011 Date of last completed: 05 April 2014
Groups:
- Xenon Including Pilot Patients: Anesthetic agent before and after CPB: xenon
- Sevoflurane: Anesthetic agent before and after CPB: sevoflurane
- TIVA: Anesthetic agent before and after CPB: propofol
Period: Overall Study
Arm/Group | Xenon Including Pilot Patients | Sevoflurane | TIVA
Started | 178 | 165 | 166
Completed | 177 | 165 | 163
Not Completed | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): randomised and treated patients
Groups:
- Xenon: Anesthetic agent before and after CPB: xenon
- Total: Total of all reporting groups
Arm/Group | Xenon | Sevoflurane | TIVA | Total
Number analyzed (Participants) | 161 | 165 | 166 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.66 (9.12) | 63.86 (8.66) | 63.89 (9.40) | 64.14 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 20 | 64
  Male | 142 | 140 | 146 | 428
Region of Enrollment [Number; unit: participants]
  Netherlands | 12 | 11 | 11 | 34
  Italy | 3 | 4 | 4 | 11
  France | 89 | 93 | 93 | 275
  Germany | 57 | 57 | 58 | 172
BMI [Mean (Standard Deviation); unit: kg/m²] | 27.65 (3.64) | 27.21 (3.68) | 27.78 (4.00) | 27.55 (3.78)

OUTCOME MEASURES:

1. Primary Outcome: Blood Level of Troponin I
Description: Blood level of troponin I measured by a central laboratory
Time Frame: Sampling performed 24 hours after the end of the surgical procedure
Population: The primary analysis was a non-inferiority comparison between Xenon and Sevoflurane and was performed on the Per Protocol (PP) Set composed of all randomised and treated patients with no major protocol deviations during the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 146 | 151
ng/mL | 2.16 [1.54 to 2.78] | 2.57 [1.96 to 3.18]
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; Test type: Non-Inferiority or Equivalence — Xenon was to be concluded non-inferior to sevoflurane if the upper bound of the 2-sided 95% CI for the difference [mean troponin I level (xenon) - mean troponin I level (sevoflurane)] was below the prespecified margin of 0.63 ng/mL. Assuming a margin of 0.63, a same concentration of troponin I at 24 hours in the xenon and sevoflurane groups, a common standard deviation of 1.9 ng/mL and a one-sided type I error of 0.025, 164 patients per group were deemed necessary to demonstrate non-inferiority; p = 0.02, ANCOVA; Treatment difference and 95%CI assessed using ANCOVA with 24h troponin I as response, treatment group and pre-induction troponin I as covariates; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.27 to 0.47]

2. Secondary Outcome: Depth of Anaesthesia
Description: On-line monitoring of depth of anaesthesia from bi-spectral electroencephalogram analysis (BIS monitor)
Time Frame: 4 hours
Reporting Status: Not Posted

3. Secondary Outcome: Arterial Oxygen Saturation
Description: Arterial blood gases
Time Frame: 4 hours
Reporting Status: Not Posted

4. Secondary Outcome: Haemodynamic Profile
Description: Monitoring of heart rate, arterial blood pressure, central venous pressure.
Time Frame: 4 hours
Reporting Status: Not Posted

5. Secondary Outcome: Presence or Absence of Postoperative Delirium
Description: Confusion Assessment Method
Time Frame: 7 days
Reporting Status: Not Posted

6. Secondary Outcome: Clinical Laboratory Tests
Time Frame: 7 days
Reporting Status: Not Posted

7. Secondary Outcome: ECG Abnormalities
Time Frame: 7 days
Reporting Status: Not Posted

8. Secondary Outcome: Vital Signs
Time Frame: 7 days
Reporting Status: Not Posted

9. Secondary Outcome: Presence of Absence of Adverse Events, Including Myocardial Infarction
Time Frame: 7 days
Reporting Status: Not Posted

10. Primary Outcome: Log-transformed Blood Level of Troponin I
Description: Blood level of troponin I measured by a central laboratory
Time Frame: Sampling performed 24 hours after the end of the surgical procedure
Population: The non-inferiority comparison between Xenon and Sevoflurane was repeated using log-transformed blood troponin levels on the PP Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Xenon | Sevoflurane
Number analyzed (Participants) | 146 | 151
ng/mL | 0.30 [0.15 to 0.44] | 0.39 [0.25 to 0.54]
Statistical Analysis 1: Comparison: Xenon vs Sevoflurane; As the residuals from the primary ANCOVA model were non-normal and skewed, the non-inferiority analysis was repeated using log-transformed blood troponin levels; Test type: Non-Inferiority or Equivalence — It was to be concluded that xenon was non-inferior to sevoflurane if the upper bound of the 2-sided 95% CI for the difference [mean troponin I level (xenon) - mean troponin I level (sevoflurane)] was below the margin of 0.15 ng/mL; p = 0.0186, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.30 to 0.11]

ADVERSE EVENTS:
Time Frame: Adverse Events observed from the start of study treatment up to 30 days.
Description: Participants at risk are the patients from the safety set
Arm/Group | Xenon Including Pilot Patients | Sevoflurane | TIVA
Serious Adverse Events (participants affected / at risk) | 30/178 | 24/165 | 26/166
Other Adverse Events (participants affected / at risk) | 154/178 | 139/165 | 143/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenon Including Pilot Patients (N=178) | Sevoflurane (N=165) | TIVA (N=166)
MYOCARDIAL INFARCTION (Cardiac disorders) | 5 (5) | 4 (4) | 3 (3)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
LOW CARDIAC OUTPUT SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
BRONCHIAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
MEDIASTINITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
SKIN INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS HAEMOPHILUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
SURGICAL SKIN TEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
POSTOPERATIVE THORACIC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
AIR EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
COMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0) | 1 (1) — General disorders and administration site conditions
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
IMPAIRED HEALING (General disorders) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
TROPONIN I INCREASED (Investigations) | 1 (1) | 0 (0) | 2 (2)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ISCHAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xenon Including Pilot Patients (N=178) | Sevoflurane (N=165) | TIVA (N=166)
Atrial fibrillation (Cardiac disorders) | 55 | 43 | 37
Tachycardia (Cardiac disorders) | 14 | 7 | 14
Bradycardia (Cardiac disorders) | 12 | 9 | 13
Pericardial effusion (Cardiac disorders) | 9 | 4 | 5
Hypotension (Vascular disorders) | 55 | 63 | 55
Hypertension (Vascular disorders) | 39 | 27 | 37
Nausea (Gastrointestinal disorders) | 23 | 19 | 18
Constipation (Gastrointestinal disorders) | 17 | 15 | 16
Vomiting (Gastrointestinal disorders) | 17 | 9 | 13
Oedema peripheral (General disorders) | 19 | 15 | 17
Pain (General disorders) | 15 | 9 | 16
Pyrexia (General disorders) | 13 | 20 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 29 | 24 | 12
Hypovolaemia (Metabolism and nutrition disorders) | 13 | 13 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 10 | 6
Electrocardiogram ST Segment Elevation (Investigations) | 18 | 22 | 13
Troponin increased (Investigations) | 10 | 13 | 11
Troponin T increased (Investigations) | 9 | 11 | 15
Bispectral index decreased (Investigations) | 9 | 0 | 0 — Bispectral index considered unexpectedly low for one investigator
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 7
Anaemia (Blood and lymphatic system disorders) | 29 | 33 | 30
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 12 | 12 | 10
Insomnia (Injury, poisoning and procedural complications) | 7 | 9 | 4
Oliguria (Renal and urinary disorders) | 19 | 17 | 15
Anxiety (Psychiatric disorders) | 9 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other